CLINICAL TRIAL: NCT03875300
Title: Best Start - Weight Management During Pregnancy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: Burdett Trust for Nursing (Other); Public Health Wales NHS Trust (Unknown); Swansea University (Other); Cardiff Metropolitan University (Other); Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CwmTUHB
Record Dates: First submitted 2019-01-28; First posted 2019-03-14 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Obesity in Pregnancy
MeSH Terms: conditions — Pregnancy in Obesity | interventions — Pregnancy

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants in the Intervention Group (Experimental): Intervention Group - will undertake a programme of 7 x 2 hour group sessions, following the scripted 'Foodwise in Pregnancy' manual of nutrition information; practical cooking sessions; and information on low impact exercise.
  Interventions: Behavioral: Foodwise in Pregnancy
- Participants in the Control Group (No Intervention): Control Group - will continue with routine antenatal care, unchanged.

INTERVENTIONS:
Behavioral: Foodwise in Pregnancy — A 7 week programme of nutrition and lifestyle advice, delivered in community venues by trained Healthy Lifestyle Support Workers (HLSWs). Participants must meet study inclusion criteria.
  Arms: Participants in the Intervention Group

SUMMARY:
The investigators know that being overweight during pregnancy increases the health risks to both mum and baby. There is good evidence that diet or exercise, or both, during pregnancy can reduce excessive weight gain. The Best Start study aims to test the theory that obese pregnant women with a Body Mass Index (BMI) of 30 or over who participate in a structured programme of nutrition and lifestyle advice (Foodwise in Pregnancy ™) will achieve the recommended weight gain during pregnancy of no less than 5kg and no more than 9.1kg.

The investigators would like to find out if pregnant women with a BMI of 30 or over who receive the Best Start intervention are more likely to effectively manage weight gain during pregnancy. To achieve this, the investigators will undertake a trial that randomly puts participants into an experimental group, or a control group, which will compare those who receive the intervention to those who continue with routine antenatal care. The investigators are aiming to recruit around 500 women during the study period. 250 will receive the Best Start intervention, and 250 will continue with routine antenatal care.

The investigators would also like to find out if women who gain the recommended weight during pregnancy have better outcomes, compared to women who gain more or less weight. To do this the investigators will look at the routine information collected during antenatal and postnatal care, for both mum and baby. To do this regardless of the group clients are randomised to, the investigators will ask for permission to look at the routine information within the participants maternity record. This information includes, weight gained during pregnancy, whether the baby is born early, the type of labour and delivery, and any complications during the pregnancy or delivery that may have resulted in the need for additional care for mum or baby.

The results of the study will be prepared for publication in scientific journals, and for presentation at scientific conferences. All participants will be able to obtain a copy of the results once they have been published and any information that could identify participants will be removed.

DETAILED DESCRIPTION:
The intervention will invite obese pregnant women with a BMI ≥30 to participate in a research study where participants may be offered a programme of nutrition and lifestyle advice, unless participants meet the exclusion criteria.

The programme of nutrition and lifestyle advice will comprise a series of weekly 7 x 2 hour group sessions, which will be delivered in community venues by trained Healthy Lifestyle Support Workers (HLSWs) employed within the maternity service.

The group sessions will follow the scripted "Foodwise in PregnancyTM" manual of nutrition information; practical cooking sessions; and information on low impact exercise e.g. walking. 'Foodwise in PregnancyTM' has been developed by a group of NHS Dietitians and Midwives and is adapted from the existing Foodwise for Life programme. Pedometers will be provided at session three to raise participants awareness of the benefits of physical activity. The programme is participative in its approach to experiential learning.

The group sessions will also promote breastfeeding (All Wales Maternity Strategy Key Performance Indicator/Measure) to assist healthy weight gain for babies, healthy weaning and the importance of play and physical activity. Delivery of the sessions will be quality assured by a specialist public health dietitian and public health midwife employed within Cwm Taf University Health Board.

Because eligible women will initially be referred by a midwife, all midwives will be trained by a public health dietitian on the "Eating for 1, Healthy and Active for 2" Royal College of Midwives accredited compact training, to ensure a sensitive and effective conversation (using motivational interviewing techniques) that raises the issue of excess weight in pregnancy. The Healthy Lifestyle Support Workers, delivering the intervention, will also attend this training.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who at their early pregnancy dating scan (optimum time 12 weeks gestation, but with a tolerance of up to 16 full weeks gestation for women who book late) have a BMI of 30 or over and reside in Cwm Taf University Health Board area.
* Aged over 16.
* Capable of giving informed consent.
* Singleton and multiple pregnancies.

Exclusion Criteria:

* Pregnant women who at their early pregnancy dating scan (optimum time 12 weeks gestation, but with a tolerance of up to 16 full weeks gestation for women who book late) have a BMI of less than 29.9 and reside in Cwm Taf University Health Board area.
* Aged under 16.
* Incapable of giving informed consent.
* Any women who have pre-existing diabetes, or develop gestational diabetes during their pregnancy.
* Any health condition that means the health professional looking after the patient feels would contra-indicate involvement in this programme (e.g. losing the ability to consent during the programme)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index - Weight and height recordings will be used to calculate BMI in kg/m^2 at 12 weeks. | 12 weeks gestation.
  Body Mass Index.
Weight of participant recorded in kg at 36 weeks. | 36 weeks gestation.
  The odds ratio of pregnant women with a BMI of ≥30 who do not gain excessive weight and achieve the optimum recommended weight gain during pregnancy of 5-9.1kg in the intervention group compared with the control group.

SECONDARY OUTCOMES:
Number of babies born Pre-term - babies born <37 weeks. | <37 weeks gestation
  Babies born to participants of the study at <37 weeks gestation.
Number of participants identified with Pre-eclampsia - New hypertension presenting after 20 weeks of pregnancy with significant proteinuria. | 20 weeks +.
  Participants will be monitored for signs of pre-eclampsia - hypertension and proteinuria.
Number of participants identified with Thromboembolism - venous thromboembolism (VTE) - deep vein thrombosis(DVT) or pulmonary embolism (PE). | Participant booking appointment to 4 weeks postpartum.
  All participants will be monitored for VTE, DVT and PE in early pregnancy and again during the intrapartum and postpartum periods.
Mode of delivery - Caesarean section. | Date of delivery.
  Participants delivering by Caesarean section will be recorded.
Post surgical site infection - a type of healthcare associated infection in which a wound infection occurs after an invasive (surgical) procedure. | Date of delivery to 4 weeks postpartum.
  Signs of post post-surgical infections will be monitored and treated.
Number of participants identified with Postpartum haemorrhage (PPH); Primary and Secondary. | 24 hours post-delivery to 12 weeks postpartum.
  Participants will be monitored for signs of PPH.
  PPH can be broken down into stages:
  Stage 1: 500-999ml blood loss; Stage 2: 1000-1499ml blood loss; Stage 3:>1500ml blood loss (major obstetric haemorrhage); Primary postpartum haemorrhage (PPH) the loss of > 500ml of blood after vaginal delivery or < 1000ml of blood after caesarean section delivery within 24 hours of delivery. Secondary PPH is defined as abnormal bleeding from the birth canal between 24 hours and 12 weeks postnatally.
Number of participants referred to the study. | July 2017-September 2018.
  Number of obese pregnant women referred into the programme by their midwife.
Number of participants Breastfeeding at birth, and exclusively breastfeeding at 10 days and 6 months. | Postnatal; Birth; 10 days and 6 months.
  The number of study participants who breastfeed at birth, and exclusively breastfeed at 10 days and 6 months.
Percentage of weight management programme sessions attended by participants. | Programme completion, an average of 7 weeks.
  Uptake and acceptability of the programme to obese pregnant women measured through the percentage of weight management programme sessions attended.
Number of post programme interviews/focus groups with eligible participants, following a scripted questionnaire. | Programme completion, an average of 7 weeks.
  Uptake and acceptability of the programme to obese pregnant women measured through the number of post study interviews/focus groups with eligible participants.
Self reported changes in study participants measured through a self completed questionnaire at the end of the weight management programme. | Programme completion, an average of 7 weeks.
  Self reported changes in nutrition knowledge, skills, physical activity levels, confidence and behaviour.
Number of low birth weight babies born, weighing < 2.5kg. | At birth.
  Weight of baby at birth lower than 2.5kg.
Number of high birth weight babies born - Macrosomia. | At birth.
  Weight of baby at birth higher than 3.99kg
Number of Stillbirths. | 24 weeks gestation to date of delivery.
  Stillbirth - Baby born dead after 24 weeks gestation.
Number of Neonatal deaths. | Date of birth to 28 days.
  Neonatal death - Death of a baby within the first 28 days of life.
Number of babies born needing Transitional Care. | From birth to 14 days postpartum.
  Babies born needing enhanced care but not Special Care Baby Unit (SCBU)admission.
Number of babies born needing Neonatal intensive care unit (NICU) admission. | From birth to 14 days postpartum.
  Babies born needing intensive care intervention.
Rate of obesity in children born to study participants at age 4-5 years. Weight and height will be combined to calculate BMI in kg/m^2. | Age 4-5 years.
  Rate of obesity measured at age 4-5 years, recorded as part of the Child Measurement Programme for Wales (All Wales Surveillance System).
Acceptability of the programme to relevant staff groups - measured through semi-structured audio recorded interview (face-to-face or via telephone). | Up to 12 months.
  The acceptability of the programme to relevant staff groups will be assessed though 1:1 or focus group sessions. A sample of healthcare professionals to include midwife, dietician, healthy lifestyle support worker, obstetrician, sonographer, anaesthetist. Open and closed ended questioning.

OTHER OUTCOMES:
Smoking status of study participant. Self reported measure and confirmed using piCObaby Smokerlyzer CO parts per million (PPM). | Through study completion, an average of 1 year.
  Self reported and CO validated measurement of study participant smoking status at initial booking interview and self-reported at 36 weeks.
Folic acid compliance of study participant. Self reported measure. Pre-conception folic acid and early pregnancy folic acid at initial booking assessment. Recorded by Midwife. | Through study completion, an average of 1 year.
  Self reported assessment confirmed and recorded by Midwife.
Socio-economic status of study participant derived from Welsh Index of Multiple Deprivation (WIMD) using Postcode. | Through study completion, an average of 1 year.
  Socio-economic status assessed from WIMD category.
Alcohol consumption status of study participant at initial booking assessment and end of pregnancy. Self reported units consumed per week. | Through study completion, an average of 1 year.
  Alcohol consumption status. At booking and end of pregnancy. Recorded by Midwife.
Substance misuse status at booking interview. Self reported recorded by Midwife. | Through study completion, an average of 1 year.
  Substance misuse status.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Jones, Principal Investigator — Public Health Wales NHS Trust; Angela Jones, Study Director — Public Health Wales NHS Trust
Locations (4):
- United Kingdom (4):
  - Royal Glamorgan Hospital, Llantrisant
  - Prince Charles Hospital, Merthyr Tydfil
  - Ysbyty Cwm Cynon Hospital, Mountain Ash
  - Ysbyty Cwm Rhondda Hospital, Tonypandy

IPD SHARING:
Plan to Share IPD: Yes
Study findings will be disseminated via The Burdett Trust for Nursing, Cwm Taf University Health Board, Public Health Wales NHS Trust, health boards and interested clinicians and submission of a paper to a scientific journal for peer-review e.g. the British Journal of Midwifery.
  The results of our study will be prepared for publication in scientific journals, and for presentation at scientific conferences. All participants will be able to obtain a copy of the results once they have been published, no patient identifiable information will be included.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It is anticipated that the initial study findings will be available for dissemination by approximately January 2021.
  The final Statistical Analysis Plan (SAP) is still to be determined.
Access Criteria: Access criteria is still to be determined.